CLINICAL TRIAL: NCT00367471
Title: A Phase I, Dose Escalation Study to Assess the Safety and Tolerability of Lapatinib in Combination With Carboplatin, Paclitaxel, With and Without Trastuzumab in Subjects With Metastatic Breast Cancer
Brief Title: Combination Of Lapatinib With Carboplatin, Paclitaxel, and With or Without Trastuzumab In Metastatic Breast Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF103892; CLAP016A2102 (Other: Novartis)
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Neoplasms, Breast
Keywords: metastatic; paclitaxel; lapatinib; trastuzumab; carboplatin; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Lapatinib; Carboplatin; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Subjects in Treatment Group A (in cohorts of three) will receive oral lapatinib QD (Days 1 to 28). Following lapatinib administration on Day 1, paclitaxel will be administered intravenously over one hour followed immediately by an IV infusion of carboplatin over not less than 15 minutes. Carboplatin will be followed by an initial loading dose of trastuzumab by 90 minute IV infusion (first dose only) with subsequent IV doses of trastuzumab to be given weekly over 30 minute infusion. Doses of paclitaxel and carboplatin will be administered weekly (Day 1, 8, and 15). Trastuzumab is administered on Day 1, 8, 15, and 22. Treatment cycles are repeated every four weeks.
  Interventions: Drug: lapatinib; Drug: carboplatin; Drug: trastuzumab; Drug: paclitaxel
- Group B (Active Comparator): Subjects in Treatment Group B (in cohorts of three) will receive oral lapatinib QD (Days 1 to 28). Following lapatinib administration on Day 1, paclitaxel will be administered intravenously over one hour followed immediately by a ≥15 minute intravenous infusion of carboplatin. Doses of paclitaxel, and carboplatin will be administered weekly (Day 1, 8, and 15) for three weeks with cycles repeated every four weeks.
  Interventions: Drug: lapatinib; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: lapatinib — Lapatinib (GW572016) is a potent small molecule, reversible inhibitor of both EGFR and ErbB2 tyrosine kinases
Drug: carboplatin — An alkylating agent used in the treatment of some cancers
Drug: trastuzumab — A monoclonal antibody that interferes with the HER2/neu receptor
  Arms: Group A
Drug: paclitaxel — A mitotic inhibitor used in cancer treatment

SUMMARY:
The purpose of this study is to determine the optimally-tolerated regimens (OTR) for lapatinib in combination with paclitaxel, carboplatin with and without trastuzumab in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion criteria:

* Subjects must have histologically- or cytologically-confirmed invasive breast cancer with Stage IV disease.
* Treatment Group A: Documentation of ErbB2 status (IHC 3+ or FISH+) in breast tumor specimens must be demonstrated before study enrollment. It is requested that archived breast tumor tissue be sent to a central laboratory for independent confirmation of ErbB2 status by FISH analysis.
* Treatment Group B: Documentation of ErbB2 status (IHC or FISH) in breast tumor specimen must be demonstrated before study enrollment. It is requested that archived breast tumor tissue be sent to a central laboratory for independent confirmation of ErbB2 status (FISH analysis).
* Subjects must be ≥18 years of age.
* Male or female
* Criteria for female subjects:

  * Non-child-bearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are post-menopausal defined as no menstruation for more than 12 months);
  * Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility.) This category includes women with oligomenorrhoea (severe), women who are perimenopausal, and young women who have begun to menstruate. These subjects must have a negative serum pregnancy test at screening and agree to one of the following:
* Complete abstinence from intercourse from two weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication; or
* Consistent and correct use of one of the following acceptable methods of birth control:
* male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject;
* implants of levonorgestrel;
* injectable progestogen;
* any intrauterine device (IUD) with a documented failure rate of less than 1% per year;
* oral contraceptives (either combined or progestogen only); or
* barrier methods, including diaphragm or condom with a spermicide.
* Able to swallow and retain oral medication.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Subjects may have measurable lesion(s) according to RECIST criteria as per protocol. Patients with metastases only to bone are also eligible for study enrollment.
* Subjects with stable CNS metastases or leptomeningeal involvement are eligible only if they are not taking oral steroids or enzyme-inducing anticonvulsants.
* Subjects that received prior radiotherapy must have completed radiotherapy treatment at least four weeks before enrollment and recovered from all treatment-related toxicities.
* Subjects must have a left ventricular ejection fraction (LVEF) ≥ 50% or ≥ lower limit of normal for the institution based on Multiple-gated Acquisition (MUGA) scan or echocardiogram (ECHO).
* Subjects must have adequate hematological, hepatic, and renal function.
* Hemoglobin of at least 9 gm/dL
* Absolute granulocyte count of at least 1,500/mm3 (1.5 x 109/L)
* Platelets of at least 100,000/mm3 (100 x 109/L)
* Total bilirubin not more than 2.5mg/dL
* ALT and/or AST not more than 1.5 times the upper limit of the normal range (ULN) and alkaline phosphatase not more than 2.5 times the ULN. For subjects with liver metastases, AST or ALT not more than 5 times the ULN may be enrolled if the total bilirubin is less than 1.5 times the ULN and if the ALT and AST is checked twice with an interval of at least 2 weeks prior to treatment to determine that liver function is stable.
* Calculated creatinine clearance (ClCr) of at least 50mL/min according to the formula of Cockcroft and Gault as per protocol.
* Subjects who received a taxane as part of adjuvant or neoadjuvant therapy are eligible if they had recurrence of their disease more than six months after completion of treatment. Subjects that received trastuzumab as part of adjuvant therapy are eligible if they had recurrence of their disease more than six months after completion of treatment.
* Subjects must provide signed written informed consent.

Exclusion criteria:

* Subject has peripheral neuropathy of Grade 2 or higher;
* Subject has had prior systemic cytotoxic chemotherapy for metastatic or locally recurrent disease. Also, any subjects with prior chemotherapy in the adjuvant or neoadjuvant setting with anthracycline or anthracenedione-containing regimens with cumulative doses of ≥ 360mg/m2 of doxorubicin, ≥ 720mg/m2 of epirubicin, or ≥ 72 mg/m2 of mitoxantrone. Patients with prior hormonal therapy(ies) are eligible.
* Subjects with prior systemic investigational drugs within the past 30 days or topical investigational drugs within the past seven days;
* Subjects with uncontrolled or symptomatic angina, arrhythmias.
* Subjects with Class II to IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Subjects with a known immediate or delayed hypersensitivity or untoward reaction to paclitaxel, trastuzumab, carboplatin, or other related compounds, or to drugs chemically related to lapatinib. These include other aminoquinazolines , such as gefitinib (Iressa), erlotinib (Tarceva), or other chemically-related compounds.
* Has malabsorption syndrome, a disease affecting gastrointestinal function, or resection of the stomach or small bowel.
* Subjects taking any prohibited medications as per protocol.
* Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-12-07 (Actual); Primary Completion 2010-12-22 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Adverse events and safety evaluations | 28 days
  * The OTR for Treatment Group A (lapatinib, paclitaxel, carboplatin, and trastuzumab) will be defined as the maximum dose level at which no more than one subject out of six experiences a dose-limiting toxicity (DLT) after completing one treatment cycle.
  * The OTR for Treatment Group B (lapatinib, paclitaxel, carboplatin) will be defined as the maximum dose level at which no more than one subject out of six experiences a DLT after completing one treatment cycle.
  * Adverse events and changes from baseline in laboratory values, Multiple-gated Acquisition (MUGA) scanning/Echocardiogram (ECHO), and vital signs will be evaluated to assess safety and tolerability.

SECONDARY OUTCOMES:
Tumor response by RECIST version 1.0 | From date of randomization until the date of first documented progression or death from any cause,whichever came first, assessed up to 48.5 months
  Tumor response is assessed using Response Evaluation Criteria In Solid Tumors (RECIST), version 1.0. RECIST has 4 response categories:
  * Complete Response (CR) = disappearance of all target and non-target lesions.
  * Partial Response (PR) = at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of diameters.
  * Progressive Disease (PD) = At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline.
  * Stable Disease (SD) = neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD.
  A CR or PR should be confirmed within 4 weeks.
Duration of Response (DOR) | From date of randomization until the date of first documented progression or death from any cause,whichever came first, assessed up to 48.5 months
  Duration of Response is defined as the time from the first documented evidence of CR or PR until the first documented sign of PD or death due to breast cancer.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or death from any cause,whichever came first, assessed up to 48.5 months
  Progression-free survival is defined as the time from first dose until the first documented sign of disease progression or death due to any cause. For subjects who do not progress or die, but who permanently discontinue Lapatinib treatment, progression-free survival will be censored at the time of last radiological scan preceding the initiation of alternative anti-cancer therapy. For subjects who do not progress or die and who complete the study, progression-free survival will be censored at the time of last radiological scan preceding the date of the study conclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No